CLINICAL TRIAL: NCT02699307
Title: Lifestyle Intervention for Adults With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Pearl G Lee, MD, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F039731
Record Dates: First submitted 2016-02-10; First posted 2016-03-04 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): OT-led counseling based on home activity pattern
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — OT led counseling

SUMMARY:
Physical activity is the cornerstone of good diabetes management, and yet effective physical activity intervention is not available. The investigators developed a lifestyle intervention based on individual's home activity patterns. The goal of the study is to test the efficacy of this intervention among older adults with diabetes. In addition to physical activity, the investigators will also assess if the intervention will improve social participation.

DETAILED DESCRIPTION:
To tailor to the needs of older adults, the investigators developed an innovative lifestyle modification intervention that incorporates rehabilitation approaches to improve the participation of physical activities (PA) among sedentary older adults with type 2 diabetes. The intervention is developed based on well-established health behavior theory (i.e., self-regulation) and the conceptual framework from the World Health Organization, with several innovations not previously investigated in this population. The intervention:

1. is tailored based on individual's unique patterns of daily PA performed within his/her environment as opposed to the total amount of PA performed in a day or a recall of activities over some time period;
2. uses an accelerometer-assisted, field-based method to address the individual's unique physical and social environment;
3. is delivered by a trained occupational therapist in brief counseling sessions, which can be easily translated into real clinical settings; and
4. addresses participation, a patient-centered outcome that is associated with quality of life but has received limited attention outside of rehabilitation research.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Has Type 2 diabetes mellitus
* Sedentary (less than 150 minutes of exercise in week)
* English-speaking
* Community living (i.e., not a nursing home resident)
* Ambulatory with or without cane or walker
* Able to operate accelerometer
* Competent to provide informed consent

Exclusion Criteria:

* Medically unstable
* Dementia diagnosis
* Currently taking any medications for memory impairment
* Currently participating in a physical activity program
* Heart attack within the past month
* Self-reported illness or condition that would impair the cooperation with the study team or the ability to complete the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06-04 (Actual); Study Completion 2017-06-04 (Actual)

PRIMARY OUTCOMES:
Change in physical activity: accelerometer counts | baseline, 18 weeks
  Change in physical activity from baseline as measured by having participants wearing an accelerometer on their wrists for one week at home at baseline and then at the end of the study.
Change in physical activity: Community Healthy Activities Model Program for Seniors (CHAMPS) survey | baseline, 18 weeks
  Change in self reported physical activities (Kcal/week) from baseline as measured by participants answering CHAMPS survey questions at baseline and at the end of the study.

SECONDARY OUTCOMES:
Change in social participation:validated questionnaires from the Patient-Reported Outcomes Measurement Information System (PROMIS) assessment center | baseline, 18 weeks
  Changes in two subdomains of participation - ability to participate and satisfaction with participation, will be assessed by participants answering surveys at the baseline and then at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Pearl G. Lee, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No